### ASSENT TO PARTICIPATE IN RESEARCH

Dartmouth College

Study title: Children's Multimedia Study

Person leading this study: Dr. Diane Gilbert-Diamond

### Why are we doing this research study?

You can participate in this study if you want to. People do research to try to find answers to questions. We are studying how children process different types of visual media, such as watching TV, texting, and using playing games on the internet.

### Why are you being asked to be in this research study?

We need many children who are between 13 and 17 years old to participate in this study. You are in this age range and can participate *if you want to*.

## What will happen during this study?

This study will take place at Dartmouth College and will last up to two hours for each visit; you will visit us three times (Visit #1 today, Visit #2 in one to three weeks, and Visit #3 in one to three weeks).

During Visits #1, #2, and #3:

- You may eat some foods.
- You may answer simple questions.
- You may play some computer games while having your eyes tracked using an eye tracker. There will not be any object placed on your eyes.
- We may measure your height and weight.
- Your parent may be in a nearby room and you can see him/her at any time.

#### In between Visits #1 and #2:

• You will be asked to wear a physical activity monitor (like a fitbit) for up to one week.

#### What are the good things that might happen in this study?

There is little chance of good things (called benefits) happening to you from being in this research study. We hope to find benefits for people in the future.

# What are the problems that might happen in this study?

We don't know any problems that might happen during this study, except for allergic food reactions. Please let us know if you have food allergies. Some problems might happen that we don't know about. It is important to let us and your parents know right away if there is anything that you don't like about the research study. Sometimes things that bother one person don't bother another person at all, so you need to let us know when something is bothering you.

### Who will be told the things we learn about you in this study?

Only the researchers will see the information collected from you. The results of the study may be shared with other scientists, but your name will not be in any report.

### Will you get any money or gifts for being in this research study?

You will receive cash or gift cards in the following amounts in the following amounts for being in this study.

- \$30 for Visit #1
- \$20 for wearing the physical activity monitor (in between Visits #1 and #2)
- \$40 for Visit #2
- \$70 for Visit #3

If you decide in the middle of the study to not participate further, you will still receive some money.

# Who should you ask if you have any questions?

If you have questions you should ask us. If you or your parents have other questions, worries, or complaints you should call the CPHS Office at Dartmouth College (603) 646-6482.

### What if you or your parent(s) don't want you to be in this study?

Your parent needs to give us permission for you to be in this study. You do not have to be in this study if you don't want to, even if your parent has already given us permission.

### What if you change your mind?

You may stop being in the study at any time. If you want to stop, just tell us so and we will stop right away. If you decide to stop, no one will be angry or upset with you. You can ask questions at any time.

| <b>Title of Study:</b> Children's Multimedia Study <b>Principal Investigator:</b> Dr. Diane Gilbert-Diamond | |
|---|---|
| If you sign your name on this page, it means that you agree You may change your mind any time for any reason. | ee to take part in this research study |
| Sign your name here if you want to be in the study | <br>Date |
| Print your name here if you want to be in the study | |
| I have explained this study to and answered questions of<br>this form. I informed the child that he or she could stop b<br>questions at any time. From my observations, the child se<br>study. | eing in the study and can ask |
| Signature of Research Team Member Obtaining Assent | Date |
| Printed Name of Research Team Member Obtaining Asse | nt |